CLINICAL TRIAL: NCT02696317
Title: Clinical Evaluation of ACUVUE® OASYS® 1-Day Daily Disposable Silicone Hydrogel Contact Lenses
Brief Title: Clinical Evaluation of ACUVUE® OASYS® 1-Day and ACUVUE® OASYS®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CLE198-P001
Record Dates: First submitted 2016-02-24; First posted 2016-03-02 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-09

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AO1D, then AO (Other): Senofilcon A contact lenses with HydraLuxe™, followed by senofilcon A contact lenses. Each product worn bilaterally (in both eyes) for 10 days in a daily wear, daily disposable modality.
  Interventions: Device: Senofilcon A contact lenses with HydraLuxe™; Device: Senofilcon A contact lenses
- AO, then AO1D (Other): Senofilcon A contact lenses, followed by senofilcon A contact lenses with HydraLuxe™. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
  Interventions: Device: Senofilcon A contact lenses with HydraLuxe™; Device: Senofilcon A contact lenses

INTERVENTIONS:
Device: Senofilcon A contact lenses with HydraLuxe™ — Contact lenses worn during Period 1 or 2, as randomized
  Other Names: ACUVUE® OASYS® 1-Day Contact Lenses with HydraLuxe™ (AO1D)
Device: Senofilcon A contact lenses — Contact lenses worn during Period 1 or 2, as randomized
  Other Names: ACUVUE® OASYS® (AO)

SUMMARY:
The purpose of this study is to evaluate the performance of two commercially-available silicone hydrogel contact lenses in normal and low humidity environments after at least 7 days of wear.

DETAILED DESCRIPTION:
After randomization to lens order, subjects attended study visits that included a 3 hour exposure to reduced humidity environment (20% relative humidity) and subsequent tear film assessments for each study lens.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form;
* Adapted, current soft silicone hydrogel daily disposable contact lens wearer during the last 2 months;
* Prescription within power range of both study contact lenses, as stated in the protocol;
* Cylinder equal or lower than -0.75 diopter (D) in both eyes;
* Willing to wear lenses every day or at least a minimum of 5 days per week, 6 hours per day;
* Willing to discontinue artificial tears and rewetting drops on the days of study visits;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Pregnant or lactating;
* Current AO1D or AO lens wearer;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2016-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Clinical Manager, GCRA Operations, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one study center located in the United Kingdom.
Pre-assignment Details: Of the 84 enrolled, 1 subject was exited as a screen failure prior to randomization. One subject was discontinued after randomization but prior to study lenses parameter optimization. This reporting group includes all subjects exposed to habitual or study lenses (82).
Groups:
- Habitual, AO1D, AO: Habitual contact lenses worn first (to understand the baseline performance in this population), followed by senofilcon A contact lenses with HydraLuxe™ in Period 1 and senofilcon A contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 10 days in a daily wear, daily disposable modality.
- Habitual, AO, AO1D: Habitual contact lenses worn first (to understand the baseline performance in this population), followed by senofilcon A contact lenses in Period 1, then senofilcon A contact lenses with HydraLuxe™ in Period 2. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
Period: Habitual, 10 Days of Wear
Arm/Group | Habitual, AO1D, AO | Habitual, AO, AO1D
Started | 42 | 40
Completed | 40 | 36
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4
Period: Period 1, 10 Days of Wear
Arm/Group | Habitual, AO1D, AO | Habitual, AO, AO1D
Started | 40 | 36
Completed | 40 | 36
Not Completed | 0 | 0
Period: Period 2, 10 Days of Wear
Arm/Group | Habitual, AO1D, AO | Habitual, AO, AO1D
Started | 40 | 36
Completed | 39 | 36
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who were exposed to any study lenses used for parameter optimization, habitual lenses, or study lenses dispensed for 10-day wear (Full Analysis Set).
Groups:
- Overall: Habitual contact lenses worn first, followed by senofilcon A contact lenses with HydraLuxe™ and senofilcon A contact lenses in Periods 1 and 2, as randomized. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
Arm/Group | Overall
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Evaporation Rate in a Normal Environment After 10 ± 3 Days of Wear (Pre RH)
Description: Tear film evaporation rate (amount of tears that evaporates over a surface area per seconds) assessment was performed using the Oregon Health Sciences University Evaporometer. Measurements were taken on both the right and left eyes after 3 hours of wear in a normal environment after 10 ± 3 days of lens wear. The temperature and humidity were measured within an air chamber around the ocular surface with the eyes opened and closed. The evaporation from the ocular surface was calculated as the difference between the evaporation rate of the skin taken during the closed eye measurement and the evaporation rate taken during the open eye measurement. The rate of evaporation was measured in g/cm2/sec for 2 humidity ranges. A higher evaporation rate can be a contributing factor to eye irritation and lens intolerance.
Time Frame: Day 10 ± 3 days, each product
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing response.
Measure: Mean (Standard Deviation); unit: 10^-7g/cm^2/s
Units Other Than Participants: Eyes
Groups:
- ACUVUE OASYS 1-DAY: Senofilcon A contact lenses with HydraLuxe™ worn bilaterally for 10 days in a daily wear, daily disposable modality
- ACUVUE OASYS: Senofilcon A contact lenses worn bilaterally for 10 days in a daily wear, daily disposable modality
Arm/Group | ACUVUE OASYS 1-DAY | ACUVUE OASYS
Number analyzed (Participants) | 76 | 75
Number analyzed (Eyes) | 152 | 150
10^-7g/cm^2/s
  25-35% Relative Humidity | 11.97 (6.447) | 10.66 (5.700)
  35-45% Relative Humidity | 8.51 (5.562) | 7.94 (5.289)

2. Secondary Outcome: Tear Film Evaporation Rate After 10 ± 3 Days of Wear and After 3 Hours Exposure to Reduced Humidity (Post RH)
Description: Tear film evaporation rate (amount of tears that evaporates over a surface area per seconds) assessment was performed using the Oregon Health Sciences University Evaporometer. Measurements were taken on both the right and left eyes after 6 hours of lens wear, including 3 hours of wear in a 20% reduced humidity environment (20% RH), after 10 ± 3 days of lens wear. The temperature and humidity were measured within an air chamber around the ocular surface with the eyes opened and closed. The evaporation from the ocular surface was calculated as the difference between the evaporation rate of the skin taken during the closed eye measurement and the evaporation rate taken during the open eye measurement. The rate of evaporation was measured in g/cm2/sec for 2 humidity ranges. A higher evaporation rate can be a contributing factor to eye irritation and lens intolerance.
Time Frame: Day 10 ± 3 days, each product
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing response.
Measure: Mean (Standard Deviation); unit: 10^-7g/cm^2/s
Units Other Than Participants: Eyes
Arm/Group | ACUVUE OASYS 1-DAY | ACUVUE OASYS
Number analyzed (Participants) | 76 | 75
Number analyzed (Eyes) | 152 | 150
10^-7g/cm^2/s
  25-35% Relative Humidity | 11.51 (5.773) | 11.72 (5.830)
  35-45% Relative Humidity | 8.78 (5.732) | 8.68 (5.352)

3. Secondary Outcome: Pre-Lens Tear Film Minimum Protected Area (MPA) in a Normal Environment After 10 ± 3 Days of Wear (Pre RH)
Description: MPA is the minimum area of the contact lens surface (expressed in %) that is protected by the tear film during the entire interblink period. Pre-lens tear film MPA was assessed in a normal environment following 3 hours of wear. Higher values indicate less dry and more eye comfort.
Time Frame: Day 10 ± 3 days, each product
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing response.
Measure: Mean (Standard Deviation); unit: percentage of contact lens surface area
Units Other Than Participants: Eyes
Arm/Group | ACUVUE OASYS 1-DAY | ACUVUE OASYS
Number analyzed (Participants) | 76 | 75
Number analyzed (Eyes) | 152 | 150
percentage of contact lens surface area | 84.64 (27.835) | 85.37 (25.634)

4. Secondary Outcome: Pre-Lens Tear Film MPA After 10 ± 3 Days of Wear and After 3 Hours Exposure to Reduced Humidity (Post RH)
Description: MPA is the minimum area of the contact lens surface (expressed in %) that is protected by the tear film during the entire interblink period. Pre-lens tear film MPA was assessed following 6 hours of wear including 3 hours in a reduced humidity environment (20% RH).. Higher values indicate less dry and more eye comfort.
Time Frame: Day 10 ± 3 days, each product
Population: Full Analysis Set. Number Analyzed is the number of eyes with non-missing response.
Measure: Mean (Standard Deviation); unit: percentage of contact lens surface area
Units Other Than Participants: Eyes
Arm/Group | ACUVUE OASYS 1-DAY | ACUVUE OASYS
Number analyzed (Participants) | 76 | 75
Number analyzed (Eyes) | 152 | 150
percentage of contact lens surface area | 94.14 (14.399) | 91.61 (20.004)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 39 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to initiation of study treatment
- Habitual Lenses: All subjects exposed to habitual contact lenses during Period 1
- ACUVUE OASYS 1-DAY: All subjects exposed to ACUVUE OASYS 1-DAY contact lenses
- ACUVUE OASYS: All subjects exposed to ACUVUE OASYS contact lenses
Arm/Group | Pre-treatment | Habitual Lenses | ACUVUE OASYS 1-DAY | ACUVUE OASYS
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/82 | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/82 | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/84 | 0/82 | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.